CLINICAL TRIAL: NCT01642095
Title: Focal Adhesion Kinase Expression in Pediatric Renal Tumors
Brief Title: Studying Biomarkers in Samples From Younger Patients With Kidney Cancer
Status: Withdrawn | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B8; NCI-2012-01987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000736805; AREN12B8; COG-AREN12B8; AREN12B8 (Other: Childrens Oncology Group); AREN12B8 (Other: CTEP)
Record Dates: First submitted 2012-07-15; First posted 2012-07-17 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2017-10

CONDITIONS: Childhood Kidney Neoplasm; Clear Cell Renal Cell Carcinoma; Congenital Mesoblastic Nephroma; Rhabdoid Tumor of the Kidney
MeSH Terms: conditions — Carcinoma, Renal Cell; Nephroma, Mesoblastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Basic science (FAK expression): Archived tumor tissue samples are analyzed for FAK expression by IHC. IHC staining is compared in normal renal tissue, Wilms tumor (routine and anaplastic), malignant rhabdoid tumor of the kidney, clear cell sarcoma of the kidney, and mesoblastic nephroma.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This laboratory study is looking into biomarkers in samples from younger patients with kidney cancer. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors find better ways to treat cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether focal adhesion kinase (FAK) is expressed and if FAK is phosphorylated in pediatric renal tumors.

OUTLINE:

Archived tumor tissue samples are analyzed for FAK expression by immunohistochemistry (IHC). IHC staining is compared in normal renal tissue, Wilms tumor (routine and anaplastic), malignant rhabdoid tumor of the kidney, clear cell sarcoma of the kidney, and mesoblastic nephroma.

ELIGIBILITY:
Inclusion Criteria:

* Formalin-fixed, paraffin-embedded tissue samples from patients diagnosed with the following renal tumors:

  * Anaplastic Wilms tumor
  * Malignant rhabdoid tumor of the kidney
  * Clear cell sarcoma of the kidney
  * Mesoblastic nephroma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2012-09-01 (Actual)

PRIMARY OUTCOMES:
FAK expression in pediatric renal tumors | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Beierle, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States